CLINICAL TRIAL: NCT01740934
Title: An Eight-Week, Multi-Site, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Trial to Evaluate the Safety, Tolerability, and Effects of Anatabloc® Crème in Subjects With Rosacea Followed by an Open-Label Extension
Brief Title: A Study to Evaluate the Safety, Tolerability, and Effects of Anatabloc® Crème in Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rock Creek Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCP-012
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Rosacea
Keywords: rosacea; anatabine; Anatabloc; dermatology
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anatabloc Cream (Active Comparator): Twice daily use of active facial cream
  Interventions: Other: Anatabloc Cream
- Placebo Cream (Placebo Comparator): Twice daily use of placebo facial cream
  Interventions: Other: Placebo Cream

INTERVENTIONS:
Other: Anatabloc Cream — subject will apply active cream topically, twice per day according to instructions
  Arms: Anatabloc Cream
Other: Placebo Cream — subject will apply placebo cream topically, twice per day according to instructions
  Arms: Placebo Cream

SUMMARY:
This is a multi-site, four-visit, eight-week, double-blind, randomized, vehicle-controlled, parallel-group study followed by an eight-week open-label extension to evaluate the safety, tolerability, and potential effects of Anatabloc Facial Cream. The secondary aim is to evaluate if Anatabloc Facial Cream improves the appearance of the skin in subjects with mild to moderate rosacea.

ELIGIBILITY:
Inclusion Criteria:

* age between 25-70 years
* diagnosed with mild to moderate rosacea

Exclusion Criteria:

* allergy or sensitivity to the study products or their components
* severe rosacea
* current use of glucocorticoids, anti-acne products, antibiotics, topical retinoids, or vasoactive drugs
* recent oral isotretinoin use
* current use of anatabine-containing supplements (ie. Anatabloc, Anatabloc Unflavored, CigRx)

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Adverse Effects | 8 to 16 weeks
  Collected information of the safety, tolerability and adverse events, and subjective experience related to the use of Anatabloc Cream by subjects

SECONDARY OUTCOMES:
Change in the appearance of the facial skin | 8 to 16 weeks
  Change measured by comparison of questionnaire and rating scores over time

CONTACTS AND LOCATIONS:
Overall Officials: M Varga, MD, Study Director — Star Scientific
Locations (3):
- United States (3):
  - Susan H. Weinkle, MD, Bradenton, Florida
  - Lupo Center for Aesthetic & General Dermatology, New Orleans, Louisiana
  - Diane Berson, MD, New York, New York